CLINICAL TRIAL: NCT01743898
Title: A Prospective Pharmacodynamic Study of Rivaroxaban Using Peak and Trough Coagulation Test Results in Patients on Therapeutic Doses of Rivaroxaban
Brief Title: A Prospective Pharmacodynamic Study of Rivaroxaban
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Suzanne J. Francart, PharmD, CPP, Pharm. D, CPP, University of North Carolina, Chapel Hill
Other Study IDs: 12-1254
Record Dates: First submitted 2012-10-07; First posted 2012-12-06 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Blood Clot
MeSH Terms: conditions — Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental: Patient taking FDA approved dose of rivaroxaban
  Interventions: Drug: Rivaroxaban
- Control Group: Patient not taking any form of anticoagulation
  Interventions: Other: no anticoagulation

INTERVENTIONS:
Drug: Rivaroxaban — Patients will continue on their Rivaroxaban dose as previously prescribed by their individual physician. No dose adjustments will be made for the purpose of this study.
  Other Names: Xarelto
  Groups: Experimental
Other: no anticoagulation
  Groups: Control Group

SUMMARY:
The ability to explain bleeding or clotting complications in patients treated with rivaroxaban remains challenging. In addition, there is limited data on how coagulation tests perform in patients treated with therapeutic doses of rivaroxaban. Predicted responses of coagulation tests to therapeutic doses of rivaroxaban may be helpful in better understanding abnormal responses to rivaroxaban. The purpose of the study is to define a therapeutic reference range for peak and trough coagulation tests in patients taking FDA approved doses of rivaroxaban and to determine which tests may be most clinically useful for monitoring rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

Person taking therapeutic dose of Rivaroxaban

Exclusion Criteria:

* CrCl < 15 mL/min
* Non-FDA approved dose based on calculated CrCl with most recent SCr
* Age < 18 years
* Inability to communicate in the English language
* Decisionally-impaired individuals
* Incarcerated
* Pregnant/Lactating (Pregnancy category: C, unevaluated effects in lactation)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients taking FDA-approved doses of rivaroxaban and control subjects not taking an anticoagulant or antiplatelet were eligible for inclusion
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Hawes, PharmD, BCPS, CPP, Study Director — Department of Family Medicine
Locations (1):
- Carolina Point II, Chapel Hill, North Carolina, United States